CLINICAL TRIAL: NCT02196909
Title: Clinical, Biological and NMR Outcome Measures Study for Hereditary Inclusion Body Myopathy Due to Mutation of UDP-N-acetylglucosamine 2-epimerase/N-acetylmannosamine Kinase Gene (GNE)
Acronym: ClinBio-GNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ClinBio-GNE
Record Dates: First submitted 2014-04-08; First posted 2014-07-22 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: HIBM
Keywords: HIBM; GNE
MeSH Terms: interventions — Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIBM patient (Active Comparator): motor function, muscle strength, NMR, 24h urine and serum collections at baseline, then annually
  Interventions: Other: motor function and strength assessment; Other: NMR assessment; Other: 24h urine and serum collection
- Controls (Active Comparator): motor function, muscle strength, 24h urine and serum collections at baseline only
  Interventions: Other: motor function and strength assessment; Other: 24h urine and serum collection

INTERVENTIONS:
Other: motor function and strength assessment
Other: NMR assessment
  Arms: HIBM patient
Other: 24h urine and serum collection

SUMMARY:
The objective of the study is to identify the best clinical and biological outcome measures for further therapeutics approaches.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age.
* Must be willing and able to provide consent.
* Must have a genetic diagnosis of HIBM, GNE myopathy, Quadriceps Sparing Myopathy (QSM), Inclusion Body Myopathy Type 2, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease.
* Must be willing and able to comply with all study requirements.
* Affiliated to or a beneficiary of a social security category
* Must take part in the HIBM-PMP UX001-CL401 study

Exclusion Criteria:

* Received ManNAc therapy or other similar substance
* Any unrelated, comorbid disease or condition that, in the view of the investigator, would interfere with study participation or would affect safety.
* Patients with specific contraindication to MRI (i.e. metallic foreign body, claustrophobia…) will be allowed to participate, but MRI will not be performed.
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Measure of changes in motor function and muscle strength assessment between 2 time points | baseline, 1 year, 2 years, 3 years
Measure of changes in NMR upper and lower limbs assessment between 2 timepoints(not for controls) | baseline, 1 year, 2 years, 3 years
24h urine and serum collection, measures at different time points | baseline, 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Myology, Paris, France